CLINICAL TRIAL: NCT02785341
Title: Adaptated Physical Activity During Chemotherapy: Evaluation of the Psychological, Physiological and Biological Impact
Acronym: APA2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: APA2-IPC 2014-010
Record Dates: First submitted 2016-05-18; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Cancer
Keywords: adapted physical activity
MeSH Terms: conditions — Neoplasms | interventions — Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate adaptated physical activity (Group A) (Other): Group A began a physical activity program for 12 consecutive weeks from inclusion in the protocol, then underwent the usual care for 12 additional weeks.
  Then to complete five evaluations with several questionnaires, and 6-minute walk test every 6 weeks (T0, T1, T2, T3 and T4) and leptin level with a blood test every 12 weeks (T0, T2 and T4).
  Interventions: Other: questionnaires every 6 weeks (T0, T1, T2, T3 and T4); Other: 6-minute walk test) every 6 weeks (T0, T1, T2, T3 and T4); Other: leptin level with a blood test every 12 weeks (T0, T2 and T4)
- Without immediate adaptated physical activity (Group B) (Other): Group B followed the usual care for 12 weeks then started the physical activity program for 12 additional weeks.
  Then to complete five evaluations with several questionnaires, and 6-minute walk test every 6 weeks (T0, T1, T2, T3 and T4) and leptin level with a blood test every 12 weeks (T0, T2 and T4).
  Interventions: Other: questionnaires every 6 weeks (T0, T1, T2, T3 and T4); Other: 6-minute walk test) every 6 weeks (T0, T1, T2, T3 and T4); Other: leptin level with a blood test every 12 weeks (T0, T2 and T4)

INTERVENTIONS:
Other: questionnaires every 6 weeks (T0, T1, T2, T3 and T4) — Questionnaire MFI 20 Questionnaire life satisfaction Scale of measurement of the positive and negative affects Questionnaire QLQ-C30 (EORTC) Questionnaire on the personal goals
Other: 6-minute walk test) every 6 weeks (T0, T1, T2, T3 and T4)
Other: leptin level with a blood test every 12 weeks (T0, T2 and T4) — blood sample

SUMMARY:
Although treatments significantly increase the life expectancy of cancer patients, their quality of life is more or less reduced. The development of supportive care, such as physical activity, is one of the tools that should be promoted to maintain quality of life and reduce treatment side effects, including fatigue.

This study was developed to understand the different biopsychosocial effects of a physical activity program carried out with patients suffering from various types of cancers, and to facilitate and improve the implementation of this type of activity in health care facilities.

Study randomized, controlled, cross-over intervention evaluating a 12-week supervised and adapted physical activity program.

Participants were assigned to one of two groups: Group A which first follows a 12-week physical activity program, then undergoes usual care for 12 additional weeks, or Group B, which continues usual care for 12 weeks (control group) and then starts the physical activity program for 12 additional weeks. Quality of life (with questionnaires for 2 groups) , well-being, fatigue, physical capacity, leptin concentration, goal setting and level of physical activity are evaluated during this protocol.

By understanding the multidimensional effects of a physical activity program for various cancer types, depending on the time of proposing the program, by evaluating the correlations among all these variables, and by evaluating long-term effects, the IPCAPA study contributes to identifying the physical activity program which will be effective, viable and feasible for all patients undergoing chemotherapy, whatever the type of cancer.

DETAILED DESCRIPTION:
Cancer is one of the leading causes of deaths in the world, with an estimated incidence of 14.1 million per year (2012) in the world, and 355,000 in France. Despite an increase in survival rates after cancer treatment, the psychological impact of the diagnosis and the aggressiveness of treatments such as chemotherapy tend to significantly decrease the quality of life of patients during and after cancer care.

Helping patients to support regular treatment is a crucial point in increasing compliance with treatment and thus increasing the cure rate, and many supportive care have been developed and implemented. Physical activity, now regarded as a non-drug therapy, provides many benefits, both in tertiary and secondary prevention during cancer treatment. Many studies have shown a decrease in mortality with physical activity during and after treatment, especially for breast, colon and prostate cancer. Regular physical activity during treatment increases patients' quality of life, for many types of cancer. The prevalence of fatigue during cancer is well described, as well as the need to effectively treat cancer related fatigue in order to enable patients to better withstand their treatment. Within the last decade, it has been pointed out that physical activity is one of the most efficient ways to combat cancer related fatigue.

From a psychological point of view, physical activity can decrease anxiety, depression and stress, and can also increase self-esteem, perceived control, and overall mental health.

Exercise physiologically increases physical capacity, strength, endurance and flexibility, and decreases physical symptoms such as pain and nausea. Biologically, physical activity often results in beneficial changes in the circulation level of adiponectin, leptin, insulin, and C-reactive protein, especially during breast, prostate and gastric cancer. Overall, physical activity during cancer treatment results in improvement in general quality of life, including mental, physical and social dimensions.

Although physical activity during cancer treatment is known to induce many benefits, depending on the cancer and the type of treatment, it is difficult to clearly investigate the effects of physical activity during cancer and how they interact or are sequential.

A better understanding of the close relationship between the psychological and physiological aspects might allow us to better understand the effects of physical activity during cancer. Exercise programs used during cancer treatment vary from one study to another in their duration, intensity and frequency. Furthermore, not all patients are included and not all types of cancers and treatment are considered.

Our study, named Institut Paoli Calmettes Adapted Physical Activity, was developed to understand the different biopsychosocial effects of a physical activity program carried out with patients suffering from various type of cancers, and to facilitate and improve the implementation of this type of activity in health care facilities.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or more,
* Performance status (WHO) ≤ 2
* Ability to participate in the IPCAPA program and medical certification of no contraindications to exercise
* Availability and willingness to participate in the IPCAPA study for the duration of the protocol
* Affiliated to a social security system
* Signed informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding woman.
* Woman with childbirth ability without effective contraception.
* Patient in emergency situations, adult subject to a measure of legal protection (major trusteeship, guardianship or ward of court), or unable to consent.
* Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons.
* Inability to practice physical activity.
* Planned surgery within 24 weeks of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Impact of physical activity on fatigue during chemotherapy | From the inclusion in the protocol until week 24
  Questionnaire MFI 20 (Multidimensional Fatigue Inventory)

SECONDARY OUTCOMES:
Physiological evaluation | From the inclusion in the protocol until week 24
  6-minute walk test
Biological evaluation | Leptin concentration realized from inclusion (week 1) then week 12 and week 24
  Leptin level with a blood test

CONTACTS AND LOCATIONS:
Overall Officials: CAPPIELLO Maria Antonietta, MD, Principal Investigator — Institut Paoli-Calmettes

REFERENCES:
- See also: Institut PAOLI-CALMETTES — http://www.institutpaolicalmettes.fr